CLINICAL TRIAL: NCT00305630
Title: Neovascular Age Related Macular Degeneration, Periocular Corticosteroids, and Photodynamic Therapy
Brief Title: Neovascular Age Related Macular Degeneration (AMD), Periocular Corticosteroids, and Photodynamic Therapy (PDT)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Oregon Health and Science University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IND 64263
Record Dates: First submitted 2006-03-20; First posted 2006-03-22 (Estimated); Last update posted 2006-03-22 (Estimated); Status verified 2006-03

CONDITIONS: Choroidal Neovascularization; Age-Related Macular Degeneration
Keywords: Corticosteroids; Triamcinolone; Photodynamic therapy; Choroidal neovascularization; Age-related macular degeneration
MeSH Terms: conditions — Choroidal Neovascularization; Macular Degeneration

INTERVENTIONS:
Drug: Periocular injection of triamcinolone acetonide 40mg

SUMMARY:
Randomized controlled clinical trial of periocular corticosteroids as adjunctive therapy to photodynamic therapy (PDT) for patients with neovascular age-related macular degeneration (AMD). Patients undergoing PDT are randomized to either a periocular corticosteroid injection with 40 mg of triamcinolone acetonide or observation just prior to PDT. Patients are followed for 6 months. Primary outcome is leakage from choroidal neovascularization (CNV) at 3 months on fluorescein angiography.

ELIGIBILITY:
Inclusion Criteria:

* Active choroidal neovascularization
* Age related macular degeneration
* Visual acuity 20/20 to 20/400

Exclusion Criteria:

* Neovascular lesion >6500 microns is greatest linear diameter
* More than one prior photodynamic therapy treatment
* Receiving systemic corticosteroids
* Intraocular pressure > 21 mm Hg or glaucoma medication use
* History of glaucoma or history of ocular hypertension

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2002-07; Study Completion 2005-11

PRIMARY OUTCOMES:
Fluorescein leakage from choroidal neovascularization on fluorescein angiography at 3 months after randomization.

SECONDARY OUTCOMES:
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Douglas A Jabs, MD, MBA, Study Chair — Johns Hopkins University; Neil M Bressler, MD, Principal Investigator — Johns Hopkins Univeristy School of Medicine; David J Wilson, MD, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Johns Hopkins Univeristy School of Medicine, Baltimore, Maryland
  - Oregon Health Science Univeristy, Portland, Oregon